CLINICAL TRIAL: NCT02955654
Title: Acceptance and Commitment Therapy in SSRI-Resistant Obsessive Compulsive Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of finacial support
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMHC-OCD-002
Record Dates: First submitted 2016-10-31; First posted 2016-11-04 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2017-04

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Acceptance and Commitment Therapy; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acceptance and commitment therapy (Experimental): Patients randomized to ACT will receive weekly 45-50 minute sessions delivered over 8 weeks by a therapist. ACT will include mindfulness,learning new methods to handle problems，acceptance of thoughts and feelings, learning to disempower thoughts and feelings, and values-based committed action.
  Interventions: Behavioral: Acceptance and commitment therapy
- Aripiprazole (Active Comparator): Patients randomized to aripiprazole group will be treated with aripiprazole at the dose of 10-20mg/day for 8 weeks.
  Interventions: Drug: Aripiprazole
- Stress management training (Other): Patients randomized to SMT group will be received 2 introductory sessions and 15 treatment sessions. SMT will include training of stress manage-ment skills, progressive muscle relaxation,positive imagery, assertiveness training, and problem solving.
  Interventions: Behavioral: Stress management training

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — Patients randomized to ACT will receive weekly 45-50 minute sessions delivered over 8 weeks by a therapist. ACT will include mindfulness,learning new methods to handle problems，acceptance of thoughts and feelings, learning to disempower thoughts and feelings, and values-based committed action.
  Arms: Acceptance and commitment therapy
Drug: Aripiprazole — Patients randomized to aripiprazole group will be treated with aripiprazole at the dose of 10-20mg/day for 8 weeks.
  Arms: Aripiprazole
Behavioral: Stress management training — Patients randomized to SMT group will be received 2 introductory sessions and 15 treatment sessions. SMT will include training of stress manage-ment skills, progressive muscle relaxation,positive imagery, assertiveness training, and problem solving.
  Arms: Stress management training

SUMMARY:
The purpose of this study is to determine whether acceptance and commitment therapy is effective in the treatment of SSRIs-resistant obsessive- compulsive disorder.

DETAILED DESCRIPTION:
The patients who were SSRI-resistant will be randomized to ACT, aripiprazole, or SMT. Independent evaluators, blind to treatment,will evaluate patients during the study.The Yale-Brown Obsessive Compulsive Scale (YBOCS)will be used to measure OCD severity.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65;
2. no less than 9 years in education;
3. a DSM-IV diagnosis of OCD
4. moderately symptomatic (Yale-Brown Obsessive Compulsive Scale score≥16)
5. received at least two kinds of SSRIs at optimal dose for more than 12 weeks An optimal dose is described as following: clomipramine hydrochloride, at least 225 mg/d;fluoxetine, at least 60 mg/d; paroxetine hydrochloride, at least 60 mg/d; sertraline hydrochloride, at least 200 mg/d; fluvoxamine, at least 250 mg/d; citalopram hydrobromide,at least 60 mg/d; and escitalopram oxalate, at least 40 mg/d.Patients who are unable to tolerate the supposed optimal doses were also eligible if at their maximally tolerated dose.

Exclusion Criteria:

1. with comorbid Axis I psychiatric disorders
2. drug abuse in the last 3 months
3. HAMD>25
4. too severe to receive ACT or evaluation
5. at high risk of suicide
6. pregnant or prepare for pregnancy
7. with somatic disorder
8. received aripiprazole(≥10mg for 8weeks) or ACT(8 times within 2 months) before
9. treated with no more than one kind of SSRI before

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale | 0,8week
  Change from baseline Y-BOCS score at 8 weeks

SECONDARY OUTCOMES:
Beck Depression Inventory | 0,8week
Acceptance and Action Questionnaire | 0,8week
Treatment Evaluation Inventory-Short Form | 0,8week
Basic life sign | 0,8week
BMI | 0,8week
Abnormal Involuntary Movement Scale | 0,8week

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, Ph.D M.D, Study Director — Shanghai Mental Health Center

IPD SHARING:
Plan to Share IPD: Undecided